CLINICAL TRIAL: NCT03506854
Title: Phase 1, Multicenter, Open-Label, Parallel Group Adaptive Pharmacokinetic Single Dose Study Of ISIS 681257 Subcutaneous Injections In Male And Female Subjects With Normal And Impaired Renal Function
Brief Title: Study of ISIS 681257 in Patients With Renal Impairment Compared to Healthy Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akcea Therapeutics (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 681257-CS12
Record Dates: First submitted 2018-04-03; First posted 2018-04-24 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal Renal Function (Experimental): Subjects with normal renal function will be matched by age (±10 years), weight (± 20%), and gender to the pooled mean values of subjects with the moderate renal impairment. Subjects will receive 1 dose of ISIS 681257.
  Interventions: Drug: ISIS 681257
- Moderate Renal Impairment (Experimental): Presence of moderate renal impairment (eGFR 30-59 mL/min/1.73m2). Subjects will receive 1 dose of ISIS 681257.
  Interventions: Drug: ISIS 681257

INTERVENTIONS:
Drug: ISIS 681257 — Xmg dose administered as a subcutaneous injection

SUMMARY:
This is a Phase 1, Multicenter, Open-Label, Parallel Group Adaptive Pharmacokinetic Single Dose Study of ISIS 681257 Subcutaneous Injections in Male And Female Subjects with Normal and Impaired Renal Function

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* BMI 18.5 to 42.0 kg/m2
* No known diseases or significant findings on physical exam (normal renal only)
* eGFR >/= 90 mL/min/1.73m2 (normal renal only)
* Clinically stable (renal impaired only)
* eGFR 30-59 mL/min/1.73m2 (renal impaired only)

Exclusion Criteria:

* Females of childbearing potential
* Conditions or disease that may interfere with study drug
* Any significant diseases
* Hypersensitivity to any drugs or similar drugs to those used in the study
* Drug dependency or abuse
* Previous exposure to other investigational drug within 28 days
* Blood donations within 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of ISIS 681257 following a single subcutaneous dose in subjects with impaired renal function relative to matched, healthy controls with normal renal function. | Day 31
  The plasma concentrations of ISIS 681257 will be measured.

SECONDARY OUTCOMES:
The incidence of adverse effects of ISIS 681257 in subjects with normal and impaired renal function. | Day 31
  The safety of ISIS 681257 will be assessed by determining adverse effects by dose. Safety results in subjects with renal impairment dosed with ISIS 681257 will be compared with those from healthy subjects dosed with ISIS 681257.
The plasma protein binding of ISIS 681257 in subjects with normal and impaired renal function. | Day 1
  Percent of ISIS 681257 bound to proteins in subjects with renal impairment dosed with ISIS 681257 will be compared with those from healthy subjects dosed with ISIS 681257.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Clinical Site, Orlando, Florida
  - Clinical Site, Knoxville, Tennessee
- Clinical Site, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milosavljevic MN, Stefanovic SM, Pejcic AV. Potential Novel RNA-Targeting Agents for Effective Lipoprotein(a) Lowering: A Systematic Assessment of the Evidence From Completed and Ongoing Developmental Clinical Trials. J Cardiovasc Pharmacol. 2023 Jul 1;82(1):1-12. doi: 10.1097/FJC.0000000000001429. PMID 37070852